CLINICAL TRIAL: NCT06262542
Title: Efficacy and Safety of Chinese Herb Medicine-Moxibustion Therapy on Chemotherapy-Induced Leukopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Armed Forces General Hospital (Other Government)
Responsible Party: Principal Investigator, Cheng Ming Huei, Principal Investigator, Taichung Armed Forces General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111016
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cancer, Chemotherapy-induced Leukopenia, Chinese Herb Medicine-moxibustion
MeSH Terms: conditions — Neoplasms | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (moxibustion and Chinese herbal medicine group) (Experimental)
  Interventions: Other: moxibustion and Chinese herbal medicine group
- Control group (sham moxibustion and placebo herbal medicine group) (Placebo Comparator)
  Interventions: Other: moxibustion and Chinese herbal medicine group

INTERVENTIONS:
Other: moxibustion and Chinese herbal medicine group — Apply 15g of Chinese herbal powder (a mixture of scientific Chinese herbs: Jiseng Shenqi Pill, Xuanfu Daizheshi Tang, and Wendi Tang mixed in a 1:1:1 ratio, mixed with water to form a paste) to the Shénquè acupoint. Then, use 3g of 80:1 moxa wool placed in a moxibustion box for moxibustion on the lower abdomen (between the Guānyuán, Zhōngjí, and Shénquè acupoints) for 1 hour, once a day, six times a week, for a total of 12 sessions.
  sham moxibustion and placebo herbal medicine group): Same acupoint frequency, but use 15g of flour instead of herbal paste and replace moxibustion with a heated nightlight for sham moxibustion.
  Other Names: sham moxibustion and placebo herbal medicine group

SUMMARY:
Cancer is the second leading cause of death globally, with an estimated 9.6 million deaths in 2018, accounting for one-sixth of total deaths. The economic burden of cancer continues to rise globally, causing significant physiological, psychological, and economic pressures on individuals, families, communities, and healthcare systems. The toxic effects of chemotherapy, such as nausea, vomiting, decreased blood cells, fatigue, etc., can impair patients' function, activities, and quality of life. Chemotherapy-induced leukopenia (CIL), particularly low white blood cell counts (48.9%), is a major concern for cancer patients.

Current conventional treatments primarily involve colony-stimulating factors (G-CSF and GM-CSF) to accelerate neutrophil recovery and regulate granulocyte production. However, G-CSF is costly and adds financial burden, and its use is restricted to cases meeting specific criteria. Additionally, rapid changes in patients' symptoms, weakness, and poor appetite may lead to swift deterioration of their condition, making it challenging to predict and prevent. Moreover, G-CSF has frequent side effects, including skin rash, liver function abnormalities, nausea, vomiting, fever, headache, fatigue, palpitations, and increased levels of ALP, LDH, and uric acid, with bone pain being the most common.

Traditional Chinese Medicine (TCM) has been a long-standing medical practice in Eastern societies and is a legally recognized healthcare option in Taiwan, covered by national health insurance. TCM includes acupuncture, moxibustion, and Chinese herbal medicine, all of which have been researched for their potential in addressing chemotherapy-induced leukopenia.

DETAILED DESCRIPTION:
Nanjing Medical University analyzed a systematic review article 7 of 14 randomized trials of traditional Chinese medicine in improving WBC count, Card-type physical function and quality of life scale (Karnofsky Performance Scale, KPS), infectious dose, and G-CSF use. According to statistics on the rate and incidence of leukopenia, it was found that CHM chemotherapy was adjusted to use western medicine plus chemotherapy. However, clinical considerations suggest that some patients with low leukocytes have poor cosmetics and are unable to meet the three-times-a-day dosage. A review of the literature found that traditional Chinese medicine powder is applied to acupoints to treat various diseases, such as primary menstrual pain 8 and chronic obstructive pulmonary disease 9 , Vomiting after general anesthesia for orthopedic surgery 10 may be treated. There are 4 articles on the Chinese Journal online using traditional Chinese medicine to treat adverse reactions after chemotherapy, including grinding traditional Chinese medicine into paste and applying it to acupoints to improve mixed leukopenia11; analysis of the correlation between traditional Chinese medicine acupoint application in the treatment of malignant tumors from 2010 to 2020 Literature, statistics on commonly used Chinese medicines, acupoints and preparation methods, found that acupoint application can improve leukopenia, constipation, vomiting and other adverse reactions in cancer patients after chemotherapy12; Chinese medicine powder mixed with petroleum jelly and applied to acupoints combined with Chinese medicine liquid injection can improve platinum Chemotherapy drugs cause vomiting, ointment, constipation, low liver function and low blood cells13; using Guilu Erxian glue patch directly improves low white blood cells and neutrophils after chemotherapy for intestinal cancer14. Therefore, local topical traditional Chinese medicine application therapy is not used for research design.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer by Western medicine doctors.
* regardless of cancer type, gender.
* aged 20 or above, experiencing WBC < 3000/μL or ANC < 1500/μL for the first time after starting chemotherapy.

Exclusion Criteria:

* Patients not suitable for moxibustion, including those with wounds at moxibustion points.
* Patients who refuse to sign the consent form.
* Minors, pregnant women, individuals with mental illnesses, those vulnerable to harm, or in disadvantaged groups.
* Patients with leukemia, where the disease itself affects changes in blood cells.
* Patients currently receiving other forms of Traditional Chinese Medicine treatment or alternative therapies that may increase white blood cell counts.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Track the number of white blood cells | 1. Baseline, before the first treatment. 2. 2 weeks after complete twelve treatment.
  Track the number of white blood cells, absolute neutrophils, in the "Complete blood count (CBC)" before and after the test.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Huei Cheng, Principal Investigator — TAICHUNG ARMED FORCED GENERAL HOSPITAL
Locations (1):
- Taichung Armed Force General Hospital, Taichung, Taiping, Taiwan

IPD SHARING:
Plan to Share IPD: No